CLINICAL TRIAL: NCT03995147
Title: Phase II Study of Pembrolizumab In Combination With R-CHOP for Patients With Untreated, High-Risk, Non-Germinal Center-Derived DLBCL
Brief Title: Pembrolizumab in Combination With Chemotherapy for Patients With Untreated B Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-0072
Record Dates: First submitted 2019-06-17; First posted 2019-06-21 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: B Cell Lymphoma; Lymphoma; Lymphoma, B-Cell; Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — pembrolizumab; R-CHOP protocol; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: R-CHOP Protocol

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered at a fixed dose of 200mg intravenously every 3 weeks in combination with R-CHOP for 6 cycles.
  Participants that respond to the combination regiment will continue to receive pembrolizumab 200 mg IV every 3 weeks for additional 35 cycles (2 years).
Drug: R-CHOP Protocol — R-CHOP chemo-immunotherapy will be administered in combination with Pembrolizumab
  Other Names: Rituximab, Cyclophosphamide, doxorubicin, vincristine, prednisone

SUMMARY:
This study will research untreated non-germinal center diffuse large B cell lymphoma and what causes the disease and the way patients respond to pembrolizumab combined with R-CHOP chemotherapy regimen (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with a histologically confirmed diagnosis of diffuse large B cell lymphoma or high-grade B cell lymphoma of a non-germinal center phenotype according to Hans criteria are eligible for enrollment in this study.
2. International Prognostic Index (IPI) score of ≥ 3, or an age-adjusted (aa) IPI score of ≥ 2.
3. A male participant must agree to use a contraception during the treatment period and for at least 120 days after the final dose of study treatment and refrain from donating sperm during this period.
4. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
6. Have measurable disease with one or more measurable lymphoma lesions ( >1.5 cm in the long axis and >1.0 cm in the short axis).
7. Patients must be able to provide an archived tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
9. Have adequate organ function. See below for adequate organ function laboratory values:

   * Hematological

     * Absolute neutrophil count (ANC) less or equal to 1000/microliter
     * Platelets less or equal to 100,000/microliters
     * Hemoglobin less or equal to 8.0/grams per decilitre
   * Renal

     * Creatinine or Measured/calculated creatinine clearance (CrCl) greater or equal to 1.5xULN or less than or equal to 30 mililiter per minute for participants with creatinine levels less than 1.5xULN
   * Hepatic

     * Total bilirubin greater than or equal to 1.5 x ULN or direct bilirubin greater than or equal to ULN for participants with total bilirubin levels less than 1.5 x ULN
     * AST (SGOT) and ALT (SGPT) greater than or equal to 2.5 x ULN (greater than or equal to 2.5 x ULN for participants with liver involvement)

Exclusion Criteria:

1. Positive urine pregnancy test within 72 hours prior to the initiation of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
3. Has received prior anti-lymphoma therapy, including radiation therapy, chemotherapy, targeted therapy, or immunotherapy.

   Note: Prior corticosteroid treatment (<10 days in duration) to alleviate lymphoma-elated symptoms is permitted.

   Note: If participant received major surgery, he or she must have recovered adequately from complications from the intervention prior to starting study treatment.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent, with the exception of short-term corticosteroid use to control lymphoma-related symptoms as outlined above) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Other exceptions may be permitted after discussion with the principal investigator.
8. Has known active CNS involvement by lymphoma.
9. Has a diagnosis of high-grade B cell lymphoma with MYC and BCL2 and/or BCL6 gene rearrangements (double hit lymphoma), primary mediastinal lymphoma, gray zone lymphoma, composite lymphoma, or previously-untreated low-grade lymphoma with disease transformation to DLBCL.
10. Has severe hypersensitivity (≥ grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection.
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive, Hepatitis B core [HBc] antibody total reactive, or HBV virus detected) or known active Hepatitis C virus infection (defined as HCV RNA is detected). Note: All patients will be screened for prior Hepatitis B exposure prior to starting therapy. Hepatitis C testing is not required.
16. Has a known history of, or active infection with tuberculosis.
17. Has a history of solid organ transplantation.
18. Has a left ventricular ejection fraction < 45%, myocardial infarction within 6 months of initiating study treatment, New York Heart Assocation class III/IV heart failure, or any uncontrolled cardiovascular conditions.
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) rate when combining pembrolizumab with R-CHOP | 24 months

SECONDARY OUTCOMES:
Complete response (CR) rate after 6 cycles of pembrolizumab in combination with R-CHOP | 18 weeks
Event free survival (EFS) rate after 6 cycles of pembrolizumab in combination with R-CHOP | 18 weeks
Overall survival (OS) rate after 6 cycles of pembrolizumab in combination with R-CHOP | 18 weeks
Number of participants with treatment related adverse events as assessed by CTCAE v 4.0 | 29 months
  Safety and tolerability of pembrolizumab in combination with R-CHOP followed by Pembrolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Kline, MD, Principal Investigator — University of Chicago Medicine
Locations (1):
- The University of Chicago, Chicago, Illinois, United States